CLINICAL TRIAL: NCT06039254
Title: A Multicenter, Non-randomized, Open-label, Parallel-controlled Study to Evaluate the Safety and Pharmacokinetics of HRS-1780 in Healthy Subjects and Subjects With Impaired Renal Function
Brief Title: Safety and Pharmacokinetics of HRS-1780 in Healthy Subjects and Subjects With Impaired Renal Function
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shandong Suncadia Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HRS-1780-102
Record Dates: First submitted 2023-08-07; First posted 2023-09-15 (Actual); Last update posted 2023-09-15 (Actual); Status verified 2023-08

CONDITIONS: Chronic Kidney Disease
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Healthy subjects group (Experimental)
  Interventions: Drug: HRS-1780
- Mild renal impairment group (Experimental)
  Interventions: Drug: HRS-1780
- Moderate renal impairment group (Experimental)
  Interventions: Drug: HRS-1780

INTERVENTIONS:
Drug: HRS-1780 — Single dose in each arm

SUMMARY:
This is a multicenter, non-randomized, open-label, parallel-controlled study. The main objective is to evaluate the safety and pharmacokinetics of HRS-1780 in subjects with mild and moderate renal impairment versus healthy subjects, and to provide a basis for dose selection of HRS-1780 in patients with chronic kidney disease.

ELIGIBILITY:
Inclusion Criteria:

- Healthy subjects：

1. Able to understand the trial procedures and possible risks, volunteers to participate in the trial, willing and able to comply with all scheduled visits and study procedures, and provides written informed consent.;
2. Male and female, 18 to 70 years of age, inclusive;
3. Body mass index (BMI) between 18.0 and 32.0 kg/m2, inclusive;
4. Normal glomerular filtration rate;
5. No clinically significant abnormalities in physical examination, vital signs, laboratory tests, 12-lead ECG, etc. at the investigator's discretion;
6. Men and WOCBP must agree to take highly effective contraceptive methods detailed in the protocol, have no plan to have a child from signing the consent form until at least one month after IP administration, and must not undertake for sperm/egg donation. Female participants should not be lactating.

Renal impairment subjects：

1. Able to understand the trial procedures and possible risks, volunteers to participate in the trial, willing and able to comply with all scheduled visits and study procedures, and provides written informed consent.;
2. Male and female, 18 to 70 years of age, inclusive;
3. Body mass index (BMI) between 18.0 and 32.0 kg/m2, inclusive;
4. Glomerular filtration rate between 30 to 89 mL/min, inclusive;
5. Except for renal impairment and related complications, no clinically significant abnormalities in physical examination, vital signs, laboratory tests, 12-lead ECG, etc. at the investigator's discretion;
6. Men and WOCBP must agree to take highly effective contraceptive methods detailed in the protocol, have no plan to have a child from signing the consent form until at least one month after IP administration, and must not undertake for sperm/egg donation. Female participants should not be lactating.

Exclusion Criteria:

- Healthy subjects：

1. Known history or suspected of being allergic to study drug or any component of it, or significant allergic reactions to other biologic products and drugs, or severe food allergies;
2. Clinically significant abnormalities in 12-Lead ECG;
3. Severe infections, injuries, or major surgeries as determined by the investigator within 3 months prior to screening, or plans to have surgeries during the study;
4. Receipt of medical devices or another investigational drug (including placebo) within 3 months or 5 half-lives, whichever is longer prior to screening, or plans to participate in another clinical study during this study;
5. Use of any prescription medicine, over-the-counter medicine, herbal remedy, or nutritional supplement within 2 weeks prior to screening;
6. Consumption of more than 14 units of alcohol per week within 6 months prior to screening, or incapable to refrain from consuming alcohol during the study, or positive alcohol breath test result;
7. Consumption of more than 5 cigarettes daily (or products with an equivalent amount of nicotine) within 3 months prior to screening, or use of any tobacco products 48 hours prior to dosing;
8. History of illicit or prescription drug abuse or addiction in the past 5 years, or illicit or prescription drug abuse within 3 months prior to screening, or positive urine drug screen;
9. Unwilling or unable to comply with the contraceptive methods detailed in this protocol;
10. Positive hepatitis B virus, hepatitis B core antibody, hepatitis C virus, human immunodeficiency virus, or syphilis at screening;
11. History or evidence of clinically significant disorders and deemed not suitable to participate in the study by the investigator within 6 months prior to screening;
12. Inability to tolerate venipuncture blood collection;
13. Any other circumstances that, in the investigator's judgment, may increase the risk to the subject, or associated with the subject's participation in and completion of the study.

Renal impairment subjects：

1. History of kidney transplant or plan to receive a kidney transplant during the trial;
2. Known history or suspected of being allergic to study drug or any component of it, or significant allergic reactions to other biologic products and drugs, or severe food allergies;
3. Clinically significant abnormalities in 12-Lead ECG;
4. Severe infections, injuries, or major surgeries as determined by the investigator within 3 months prior to screening, or plans to have surgeries during the study;
5. Receipt of medical devices or another investigational drug (including placebo) within 3 months or 5 half-lives, whichever is longer prior to screening, or plans to participate in another clinical study during this study;
6. Except for treatment of renal impairment and related complications, use of other prescription medicine, over-the-counter medicine, herbal remedy, or nutritional supplement within 2 weeks prior to screening;
7. Consumption of more than 14 units of alcohol per week within 6 months prior to screening, or incapable to refrain from consuming alcohol during the study, or positive alcohol breath test result;
8. Consumption of more than 5 cigarettes daily (or products with an equivalent amount of nicotine) within 3 months prior to screening, or use of any tobacco products 48 hours prior to dosing;
9. History of illicit or prescription drug abuse or addiction in the past 5 years, or illicit or prescription drug abuse within 3 months prior to screening, or positive urine drug screen;
10. Unwilling or unable to comply with the contraceptive methods detailed in this protocol;
11. Positive hepatitis B virus, hepatitis B core antibody, hepatitis C virus, human immunodeficiency virus, or syphilis at screening;
12. History or evidence of clinically significant disorders and deemed not suitable to participate in the study by the investigator within 6 months prior to screening;
13. Inability to tolerate venipuncture blood collection;
14. Any other circumstances that, in the investigator's judgment, may increase the risk to the subject, or associated with the subject's participation in and completion of the study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 27 (Estimated)
Dates: Start 2023-09 (Estimated); Primary Completion 2023-11-30 (Estimated); Study Completion 2023-12-08 (Estimated)

PRIMARY OUTCOMES:
Pharmacokinetics-Cmax | Start of Treatment to end of study (approximately 1 week)
  Maximum observed concentration of HRS-1780
Pharmacokinetics-AUC0-last | Start of Treatment to end of study (approximately 1 week)
  Area under the concentration-time curve from time 0 to last time point after HRS-1780 administration
Pharmacokinetics-AUC0-inf | Start of Treatment to end of study (approximately 1 week)
  Area under the concentration-time curve from time 0 to infinity after HRS-1780 administration

SECONDARY OUTCOMES:
Pharmacokinetics-Tmax | Start of Treatment to end of study (approximately 1 week)
  Time to Cmax of HRS-1780
Pharmacokinetics-t1/2 | Start of Treatment to end of study (approximately 1 week）
  Terminal elimination half-life of HRS-1780
Pharmacokinetics-CL/F | Start of Treatment to end of study (approximately 1 week)
  Apparent clearance of HRS-1780
Pharmacokinetics-Vz/F | Start of Treatment to end of study (approximately 1 week)
  Apparent volume of distribution during terminal phase of HRS-1780
Pharmacokinetics-Cumulative excretion (Ae) | Start of Treatment to end of study (approximately 1 week)
  Cumulative amount of HRS-1780 excreted in urine
Pharmacokinetics-Cumulative excretion rate (Ae%) | Start of Treatment to end of study (approximately 1 week)
  Cumulative percentage of HRS-1780 recovered in urine
Pharmacokinetics-Renal clearance (CLr) | Start of Treatment to end of study (approximately 1 week)
  Clearance of HRS-1780 by kidney
Binding rates of plasma protein (BRPP) of HRS-1780 | Start of Treatment to end of study (approximately 1 week)
  Binding rates of plasma protein
Adverse events | Start of Treatment to end of study (approximately 1 week)
  Incidence and severity of adverse events

IPD SHARING:
Plan to Share IPD: Undecided